CLINICAL TRIAL: NCT00361517
Title: Using Serum Galactomannan Levels in a Prospective, Randomised, Non-blinded Trial to Guide Early Anti-fungal Therapy in Haematology Patients at Risk of Invasive Aspergillosis.
Brief Title: To Determine Whether Galactomannan Test Will Help to Detect Fungal Infections Early and Hence Start Treatment Early
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Dr Tan Ban Hock, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NMRC/0984/2005; IRB #291/2005
Record Dates: First submitted 2006-08-06; First posted 2006-08-08 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Aspergillosis
Keywords: GM monitoring; Immunocompromised; hematological disorder; Allogenic HSCT recipients; Aspergillus PCR assay
MeSH Terms: conditions — Aspergillosis; Hematologic Diseases | interventions — Blood Specimen Collection; amphotericin B, deoxycholate drug combination; Amphotericin B; liposomal amphotericin B; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GM test (Experimental): Twice weekly blood draws from the patients in this arm for serial GM monitoring. They will be given standard antifungal prophylaxis but no antifungal therapy unless two consecutive GM readings are positive.
  Interventions: Behavioral: Galactomannan antigen monitoring, Aspergillus PCR; Other: blood draws; Other: blood draws for GM monitoring; Drug: Amphotericin-B deoxycholate; Other: blood test
- no GM monitoring (No Intervention): in this arm the patients will not have any GM monitoring and they will be given standard antifungal prophylaxis and treatment according to the published guidelines.

INTERVENTIONS:
Behavioral: Galactomannan antigen monitoring, Aspergillus PCR — There will be blood draws twice weekly for monitoring GM antigen and once a week for Aspergillus PCR.
  Arms: GM test
Other: blood draws — Blood is drawn for monitoring of Galactomannan antigen in the blood
  Arms: GM test
Other: blood draws for GM monitoring — blood samples will be taken twice weekly for monitoring of GM antigen levels in the blood and once a week for Aspergillus PCR.
  Arms: GM test
Drug: Amphotericin-B deoxycholate — 1-1.5mg/kg, i.v, once a day
  Other Names: Fungizone, Abelcet, AmBisome, Fungisome, Amphocil,
  Arms: GM test
Other: blood test — Blood will be tested twice a week for the presence of Galactomannan.
  Arms: GM test
Other: Blood test — Blood will be drawn twice a week and it will be tested for the presence of GM(a component of the cell wall of the mold Aspergillus which is released during growth)
  Arms: GM test

SUMMARY:
Chemotherapy lowers the white blood cell count or weakens the immune system for a long time. This puts the patients at a high risk of getting a serious fungal infection of the internal organs or blood. One of these infections is caused by a mold called Aspergillus and can be life threatening. Usually doctors give preventive antifungal therapy to try to lower the risk of this infection. Despite this, patients are still at risk of getting fungal infection. This study is thus designed to test Galactomannan - a component of cell wall of Aspergillus and hence detect and treat fungal infection early.

DETAILED DESCRIPTION:
The diagnosis of invasive Aspergillosis (IA) remains a challenge in the febrile neutropenic and the hematopoietic stem cell transplant (HSCT) recipients. Recent studies have shown that early diagnosis of IA is possible in this group of high-risk patients. Serial screening of circulating Galactomannan (GM), an epitopic determinant of several antigens secreted by the Aspergillus early in its growth, has been shown to be sensitive and specific in the diagnosis of IA. This test may help us to detect IA early, thereby permitting a pre-emptive strategy to be initiated in high-risk patients. In a prospective, randomized, non-blinded study, we seek to compare the outcome of a novel GM-guided anti-fungal strategy against the conventional empirical antifungal therapy. Patients randomized to the conventional arm will not undergo serial GM monitoring, but will receive standard anti-fungal prophylaxis and standard empirical antifungal therapy in accordance with published guidelines. Patients randomized to the GM arm will receive standard anti-fungal prophylaxis but will not receive empiric anti-fungal therapy unless 2 GM readings are positive. The study aims to determine if such a strategy permits targeted, pre-emptive therapy in those at greatest risk, and spare febrile patients without evidence of fungal infection other than prolonged fever from unnecessary and potentially toxic therapy. It also aims to determine if GM guided pre-emptive antifungal therapy using Amphotericin-B deoxycholate prevents the development of proven or probable invasive aspergillosis (IA). The study will also prospectively evaluate (in a blinded fashion) the use of realtime polymerase chain reaction (RT PCR) assay in the same cohort of patients receiving GM serial monitoring, and investigate its role in the diagnosis and treatment monitoring of invasive Aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed acute leukemia or high risk myelodysplastic syndrome (MDS) receiving induction chemotherapy with expected duration of neutropenia (absolute neutrophil count of < 500/mL) of at least 10 days
2. Patients with relapsed acute leukemia or MDS receiving salvage chemotherapy with expected duration of neutropenia (absolute neutrophil count of < 500/mL) of at least 10 days
3. Patients with severe aplastic anemia (SAA) receiving chemotherapy or immunosuppressive therapy using antithymocyte globulin
4. Patients receiving allogeneic/autologous hematopoeitic stem cell transplant (HSCT) using myeloablative conditioning regimens
5. Patients are at least 12 years of age, with Karnofsky score of 70%.?
6. Patients on consolidation chemo regimens like HIDAC and HyperCVAD type B with expected duration of neutropenia (ANC < 500/ml) of at least 10 days

Exclusion Criteria:

1. Patients who are human immunodeficiency virus (HIV) infected
2. Patients with uncontrolled bacteremia or active pulmonary infection at the time of randomisation
3. Patients with pre-existing proven and probable invasive fungal infections, according to the definitions of the invasive Fungal Infections Cooperative Group of the European Organization for Research and Treatment of Cancer; Mycoses Study Group of the National Institute of Allergy and Infectious Disease [10].
4. Patients receiving concomitant piperacillin/tazobactam or co-amoxyclavulinic acid
5. Patients on palliative chemotherapy
6. Patients with history of allergy to triazoles
7. Patients with prior history of anaphylactic reaction to conventional amphotericin B
8. Patients with serum levels of aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, or bilirubin more than 5 times the upper limit of normal or renal impairment with calculated creatinine clearance < 30ml/min
9. Patients with expected life-expectancy < 72 hours

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-06-01; Primary Completion 2007-10-30 (Actual); Study Completion 2009-06-30 (Actual)

PRIMARY OUTCOMES:
Development of proven or probable invasive fungal infection, fungal related mortality and overall survival in an intention to treat basis. | During neutropenia, or, in HSCT patients, while under immunosuppressive therapy

SECONDARY OUTCOMES:
Duration of antifungal therapy and toxicity associated with antifungal therapy. | while patient is on follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ban H Tan, Dr, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Lin SJ, Schranz J, Teutsch SM. Aspergillosis case-fatality rate: systematic review of the literature. Clin Infect Dis. 2001 Feb 1;32(3):358-66. doi: 10.1086/318483. Epub 2001 Jan 26. PMID 11170942
- [Derived] Tan BH, Low JG, Chlebicka NL, Kurup A, Cheah FK, Lin RT, Goh YT, Wong GC. Galactomannan-guided preemptive vs. empirical antifungals in the persistently febrile neutropenic patient: a prospective randomized study. Int J Infect Dis. 2011 May;15(5):e350-6. doi: 10.1016/j.ijid.2011.01.011. Epub 2011 Mar 11. PMID 21397541